CLINICAL TRIAL: NCT01880008
Title: An Exploratory Study of Quantitative [18F]FLT-PET and Advanced MRI as Early Indicators of Treatment Response and Molecular Markers for Cell Proliferation in Patients With Glioblastoma Following Subtotal Resection
Brief Title: Evaluation of FLT PET and MRI as Imaging Biomarkers of Early Treatment Response in Patients With Glioblastoma
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Delphine L. Chen, MD, Assistant Professor of Radiology, Washington University School of Medicine
Other Study IDs: 08-0073
Record Dates: First submitted 2010-07-30; First posted 2013-06-18 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Glioblastoma
Keywords: positron emission tomography; magnetic resonance imaging; diffusion magnetic resonance imaging; radionuclide imaging; disease management; radiation therapy
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment: All patients included in this study were treated with temozolomide and radiotherapy after subtotal resection of a WHO grade III or IV glioma.

SUMMARY:
Glioblastoma is the most common primary malignant neoplasm of the adult brain. Even after multimodal therapy, outcomes remain poor, with a median survival of one year. Although advanced imaging methods have been suggested as molecular markers of prognosis and therapeutic response, these methods have not been validated for clinical use. In this exploratory, imaging-based, trial, thirty patients with a pathological diagnosis of glioblastoma will be followed prospectively for two years. The study examines how PET and MR imaging signals change following administration of a standard radio-chemotherapy treatment regimen to determine whether these imaging modalities can provide early indicators of response to therapeutic intervention. The investigators hypothesize that decreases in uptake of an investigational 18F-FLT PET tracer following treatment with radiation and chemotherapy will be a reliable predictor of glioblastoma response. In a more exploratory fashion, the investigators also will identify changes in diffusion and hypoxia MR imaging that may also correlate well with treatment response.

DETAILED DESCRIPTION:
Patients with glioblastoma will be imaged with FLT PET/CT followed by MRI. The FLT uptake will be correlated with advanced MRI markers of tumor progression to determine the ability of using FLT PET and MRI for predicting response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (> 18 yo) with a pathological diagnosis of malignant glioma (WHO grades III and IV, including all histological subtypes)
* Surgical intervention includes subtotal resection or biopsy with MRI evidence of residual disease after resection
* Patients with plan to undergo standard chemotherapy and radiation protocols including a combination of fractionated radiation and temozolomide
* Preoperative Karnofsky performance score (KPS) of > 60
* Willingness of patient and his/her partner to use contraceptive measures for duration of trial that will include PET studies.

Exclusion Criteria:

* Patient refuses adjunctive therapy
* Pregnancy
* Karnofsky scale < 60
* Inability to undergo MR imaging studies
* Estimated GFR ≤ 60 ml/min (using GFR = 0.85*[140 - age(y)]*[bodyweight(kg)]/[72*Cr(mg/dl)] for women and GFR = [140 - age(y)]*[bodyweight(kg)]/[72*Cr(mg/dl)] for men).
* Inability or unwillingness to follow instructions for both PET and MR imaging sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with WHO grade III or IV glioma
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2008-04; Primary Completion 2010-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in FLT uptake, measured by SUV tumor/SUV normal contralateral white matter | Before and after chemotherapy/radiation therapy
  Determines the change in FLT uptake as a result of chemotherapy/radiation therapy

SECONDARY OUTCOMES:
Survival | 2 years
  Number of months from date of diagnosis to date of death.
Ki-67 | At diagnosis
  Ki-67 proliferation index on tumor specimens obtained at biopsy or from surgical resection specimen
Radiographic progression defined by MacDonald criteria | 2 years
  MacDonald criteria to be used to determine whether tumor progress or not during the course of this study
O(6)-methylguanine DNA-methyltransferase (MGMT) activity | prior to treatment
  MGMT activity from tumor specimens
Time to progression | 2 years
  Months after completing radiation treatment to first instance of radiographic progression

CONTACTS AND LOCATIONS:
Overall Officials: Delphine L Chen, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Barnes-Jewish Hospital, St Louis, Missouri, United States